CLINICAL TRIAL: NCT00555763
Title: Assessment of a New Goldmann Applanation Tonometer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Haag-Streit AG (Industry)
Responsible Party: Milko Iliev, MD, University Hospital Inselspital; Berne
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1410; 162/07
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Intraocular Pressure
Keywords: Intraocular pressure; Goldmann tonometry; applanation tonometry; Tonometry, Ocular
MeSH Terms: interventions — Manometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Device: Tonometry

INTERVENTIONS:
Device: Tonometry — Tonometry : measurement of intraocular pressure with an applanation tonometer

SUMMARY:
The classic Goldmann applanation tonometer has been further developed. The applanation principle has been retained, while the internal force transmission and the pressure gauging have been optimized, and the display of results digitized.

The purpose of the study is to compare the standard Goldmann applanation tonometer AT900 with the new version of the device, and to test the reliability and reproducibility of measurements, as well as its safety.

DETAILED DESCRIPTION:
The classic Goldmann applanation tonometer has been further developed. The applanation principle has been retained, while the internal force transmission and the pressure gauging have been optimized, and the display of results digitized.

The purpose of the study is to compare the standard Goldmann applanation tonometer AT900 with the new version of the device, and to test the reliability and reproducibility of measurements, as well as its safety.

Patients at the Department of Ophthalmology, University of Bern, will be included after informed consent. The study has been approved by the local ethical committee. Routine ophthalmologic examination will be performed and inclusion criteria evaluated. Measurements will be taken with the two tonometers in random order. Prior to pressure measurement, central corneal thickness will be measured with a non-contact method (Optical Low Coherence Reflectometry, OLCR pachymeter, Haag-Streit, Koeniz, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* patient willing to participate and signed informed consent

Exclusion Criteria:

* patient under 18 y of age
* patient pregnant
* not steady fixation, nystagm
* corneal scars or corneal disease
* astigmatism higher than 2.5 diopters
* corneal surgery in the past
* microphthalmos or buphthalmos
* contact lens wear
* dry eye syndrome
* blepharospasm
* active inflammation of conjunctiva, cornea or uvea
* known allergy to topical oxybuprocain for topical anaesthesia
* known allergy to fluorescein solution (used for applanation tonometry)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure in mmHG | single event

SECONDARY OUTCOMES:
safety of measurement | single event, up to one week post measurement

CONTACTS AND LOCATIONS:
Overall Officials: Milko E Iliev, MD, Principal Investigator — University Eye Hospital Berne; Sebastian Wolf, MD, Study Director — University Eye Hospital Berne
Locations (1):
- University Eye Hospital Berne, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] SCHMIDT TA. The clinical application of the Goldmann applanation tonometer. Am J Ophthalmol. 1960 May;49:967-78. doi: 10.1016/0002-9394(60)91818-3. No abstract available. PMID 14443098
- [Background] GOLDMANN H, SCHMIDT T. [Further contribution to applanation tonometry]. Ophthalmologica. 1961 Jun;141:441-56. doi: 10.1159/000304099. No abstract available. German. PMID 13706587
- [Background] GOLDMANN H, SCHMIDT T. [Applanation tonometry]. Ophthalmologica. 1957 Oct;134(4):221-42. doi: 10.1159/000303213. No abstract available. German. PMID 13484216